CLINICAL TRIAL: NCT05175170
Title: Fertility Decision-Making in Youth and Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Diane Chen, Behavioral Health Director; Associate Professor of Psychiatry and Behavioral Sciences, & Pediatrics, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 5R21HD097459 (NIH)
Record Dates: First submitted 2021-12-02; First posted 2022-01-03 (Actual); Results first posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Transgender Adolescents & Young Adults
Keywords: fertility; decision-making
MeSH Terms: interventions — Decision Support Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Decision-aid (Experimental): Participants will spend up to one hour freely navigating the web-based decision aid. They will complete pre- and post-test measures to determine if using the decision-aid website increased knowledge and impacted decision self-efficacy regarding fertility and fertility preservation.
  Interventions: Behavioral: Decision-aid

INTERVENTIONS:
Behavioral: Decision-aid — The decision aid consists of domains related to human reproduction, fertility, and fertility preservation. The domains address priority learning objectives in each domain to increase knowledge on the impact of gender-affirming medical interventions on fertility and fertility preservation options.

SUMMARY:
The aim of this study is to test if using a web-based medical decision-making tool on the topics of fertility and fertility-preservation increases knowledge among transgender youth and young adults.

DETAILED DESCRIPTION:
The pilot trial of Aid for Fertility-Related Medical Decisions (AFFRMED) is a single-arm, pre-/post- feasibility, acceptability, and preliminary efficacy trial. 10 transgender adolescents and young adults (AYA) and 10 parents of transgender AYA participated in a 90-120 min, virtual research visit via Zoom. During this visit they completed pre-test measures of fertility knowledge and decisional self-efficacy, followed by up to 1 hour to freely navigate AFFRMED decision aid. After using AFFRMED, participants completed post-test measures of fertility knowledge and decisional self-efficacy, as well as implementation outcomes measures (Acceptability of Intervention, Intervention Appropriateness Measure, and Feasibility of Intervention Measure).

ELIGIBILITY:
Inclusion Criteria:

* (1) youth is between the ages of 8-14 years
* (2) youth self-asserts a transgender identity
* (3) youth has expressed interest in GnRHa or is currently on GnRHa treatment; or
* (1) AYA is between the ages of 13-24 years,
* (2) AYA self-asserts a transgender identity, and
* (3) AYA has expressed interest in gender-affirming hormone (GAH) or is currently on GAH treatment.
* Parents of eligible youth will be eligible to participate.

Exclusion Criteria:

* (1) youth/parents are unable to read, speak or understand English
* (2) youth/parents are unable or unwilling to provide consent/assent/parental permission for study participation.

Ages: 8 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Youth and young adults who identify as transgender, trans, nonbinary, gender fluid, or genderqueer
Enrollment: 20 (Actual)
Dates: Start 2021-06-03 (Actual); Primary Completion 2021-10-09 (Actual); Study Completion 2021-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diane Chen, PhD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Transgender Youth and Young Adults: Transgender youth and young adults will navigate the decision-aid consisting of domains related to human reproduction, fertility, and fertility preservation. The domains address priority learning objectives in each domain to increase knowledge on the impact of gender-affirming medical interventions on fertility and fertility preservation options.
- Parents of Transgender Youth and Young Adults: Parents of transgender youth and young adults will navigate the decision-aid consisting of domains related to human reproduction, fertility, and fertility preservation. The domains address priority learning objectives in each domain to increase knowledge on the impact of gender-affirming medical interventions on fertility and fertility preservation options.
Period: Overall Study
Arm/Group | Transgender Youth and Young Adults | Parents of Transgender Youth and Young Adults
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Transgender Youth and Young Adults | Parents of Transgender Youth and Young Adults | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.5 (3.779) | 45.00 (4.83) | 30.25 (15.711)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 3 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 8 | 10 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 6 | 8 | 14
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Fertility-related Knowledge
Description: The primary study outcome is change in fertility-related knowledge from same-day pre-AFFRMED to post-AFFRMED exposure. Participants will complete a fertility-related knowledge test instrument immediately prior to AFFRMED exposure. Participants will be given 1 hour to freely navigate the web-based AFFRMED prototype. Thereafter, participants will get a 5-minute break before completing a post-AFFRMED fertility knowledge test. The knowledge test consists of 41 items, and reflects a percentage correct score ranging from 0-100% correct.
  The Mean Difference results reflect the difference in fertility knowledge test mean scores between pre-AFFRMED and post-AFFRMED exposure.
Time Frame: Pre-treatment and immediately post-treatment (same day)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transgender Youth and Young Adults | Parents of Transgender Youth and Young Adults
Number analyzed (Participants) | 10 | 10
score on a scale
  Pre-test Score | 51.463 (21.585) | 67.073 (6.729)
  Post-test Score | 85.366 (14.858) | 93.171 (2.998)
Statistical Analysis 1: Comparison: Transgender Youth and Young Adults; The hypothesis of this analysis was that using the AFFRMED would increase fertility-related knowledge. This paired-samples t-test compares participants' pre- and post-test knowledge scores; Test type: Other; p < .001, t-test, 1 sided; Mean Difference (Final Values) = -33.902
Statistical Analysis 2: Comparison: Parents of Transgender Youth and Young Adults; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < .001, t-test, 1 sided; Mean Difference (Final Values) = -26.098

2. Secondary Outcome: Change in Decisional Self-Efficacy
Description: The secondary study outcome is change in decisional self-efficacy for fertility-related decision-making from same-day pre-AFFRMED to post-AFFRMED exposure using the Decision Self Efficacy Scale. Decision Self Efficacy Scale scores range from 0 [not at all confident] to 100 [very confident]. A score of 0 indicates 'extremely low self-efficacy' and a score of 100 indicates 'extremely high self-efficacy'.
  The Mean Difference results reflect the difference in decisional self-efficacy mean scores between pre-AFFRMED and post-AFFRMED exposure.
Time Frame: Pre-treatment and immediately post-treatment (same day)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transgender Youth and Young Adults | Parents of Transgender Youth and Young Adults
Number analyzed (Participants) | 10 | 10
score on a scale
  Pre-test Score | 61.364 (17.309) | 83.864 (15.653)
  Post-test Score | 80.303 (14.903) | 92.929 (9.739)
Statistical Analysis 1: Comparison: Transgender Youth and Young Adults; The hypothesis of this analysis was that using the AFFRMED would increase fertility-related decision self-efficacy. This paired-samples t-test compares participants' pre- and post-test decision self-efficacy scores; Test type: Other; p = 0.002, t-test, 1 sided; Mean Difference (Final Values) = -20.202
Statistical Analysis 2: Comparison: Parents of Transgender Youth and Young Adults; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.051, t-test, 1 sided; Mean Difference (Final Values) = -8.081

3. Other Pre Specified Outcome: Participant-Reported Feasibility of AFFRMED
Description: The other study outcomes are related to participant-reported feasibility of the AFFRMED. Participants will also be asked to rate the feasibility of the AFFRMED using the validated Feasibility of Intervention Measure (FIM). Scale scores range from 4 to 20, with higher scores indicating greater feasibility.
Time Frame: Immediately post-treatment (same day)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transgender Youth and Young Adults | Parents of Transgender Youth and Young Adults
Number analyzed (Participants) | 10 | 10
score on a scale | 17.50 (3.308) | 18.60 (2.366)

4. Other Pre Specified Outcome: Participant-Reported Acceptability of AFFRMED
Description: The other study outcomes are related to participant-reported acceptability of the AFFRMED. Participants will also be asked to rate the acceptability of the AFFRMED using the validated Acceptability of Intervention Measure (AIM). Scale scores range from 4 to 20, with higher scores indicating greater acceptability.
Time Frame: Immediately post-treatment (same day)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transgender Youth and Young Adults | Parents of Transgender Youth and Young Adults
Number analyzed (Participants) | 10 | 10
score on a scale | 16.70 (4.244) | 18.90 (1.853)

5. Other Pre Specified Outcome: Participant-Reported Appropriateness of AFFRMED
Description: The other study outcomes are related to participant-reported appropriateness of the AFFRMED. Participants will also be asked to rate the appropriateness of the AFFRMED using the validated Intervention Appropriateness Measure (IAM). Scale scores range from 4 to 20, with higher scores indicating greater appropriateness.
Time Frame: Immediately post-treatment (same day)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transgender Youth and Young Adults | Parents of Transgender Youth and Young Adults
Number analyzed (Participants) | 10 | 10
score on a scale | 17.30 (3.917) | 18.20 (3.011)

ADVERSE EVENTS:
Time Frame: 2 hours
Arm/Group | Transgender Youth and Young Adults | Parents of Transgender Youth and Young Adults
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-02-25): https://cdn.clinicaltrials.gov/large-docs/70/NCT05175170/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-07): https://cdn.clinicaltrials.gov/large-docs/70/NCT05175170/SAP_001.pdf